CLINICAL TRIAL: NCT05230368
Title: A Pilot Open Label Phase I Trial to Evaluate the Safety and the Tolerability of a Combination of Two HIV-1 Inducers in HIV+ Sub-type B Patients Under cART With Undetectable Viral Load
Brief Title: Evaluation of the Safety and the Tolerability of a Combination of Two HIV Inducers in Patients With Undetectable Viral Load
Acronym: SYNACTHIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: INSERM SC10-US19 (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 171 SYNACTHIV
Record Dates: First submitted 2021-12-23; First posted 2022-02-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: HIV-1-infection, Subtype b

STUDY DESIGN:
Intervention Model Description: This is a monocenter pilot open label phase I trial. This trial will evaluate new procedures in LRA administration in 3 successive cohorts of 5 patients each receiving 1, 2 and 4 cycles respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1 cycle of treatment (Cohort 1 = 5 patients) (Experimental): * decitabine (5mg/m²) at days 1, 2, 3
  * romidepsin (5mg/m²) at days 4, 11, 18
  Interventions: Drug: Decitabine cycle 1; Drug: Romidepsin cycle 1
- 2 cycles of treatment (Cohort 2 = 5 patients) (Experimental): * decitabine (5mg/m²) at days 1, 2, 3, 35, 36, 37
  * romidepsin (5mg/m²) at days 4, 11, 18, 38, 45, 52
  Interventions: Drug: Decitabine cycle 1; Drug: Romidepsin cycle 1; Drug: Decitabine cycle 2; Drug: Romidepsin cycle 2
- 4 cycles of treatment (Cohort 3 = 5 patients) (Experimental): * decitabine (5mg/m²) at days 1, 2, 3, 35, 36, 37, 70, 71, 72, 105, 106, 107
  * romidepsin (5mg/m²) at days 4, 11, 18, 38, 45, 52, 73, 80, 87, 108, 115, 122
  Interventions: Drug: Decitabine cycle 1; Drug: Romidepsin cycle 1; Drug: Decitabine cycle 2; Drug: Romidepsin cycle 2; Drug: Decitabine cycle 3; Drug: Romidepsin cycle 3; Drug: Decitabine cycle 4; Drug: Romidepsin cycle 4

INTERVENTIONS:
Drug: Decitabine cycle 1 — Decitabine administration (5mg/m²) at days 1, 2, 3
Drug: Romidepsin cycle 1 — Romidepsin administration (5mg/m²) at days 4, 11, 18
Drug: Decitabine cycle 2 — Decitabine administration (5mg/m²) at days 35, 36, 37
  Arms: 2 cycles of treatment (Cohort 2 = 5 patients); 4 cycles of treatment (Cohort 3 = 5 patients)
Drug: Romidepsin cycle 2 — Romidepsin administration (5mg/m²) at days 38, 45, 52
  Arms: 2 cycles of treatment (Cohort 2 = 5 patients); 4 cycles of treatment (Cohort 3 = 5 patients)
Drug: Decitabine cycle 3 — Decitabine administration (5mg/m²) at days 70, 71, 72
  Arms: 4 cycles of treatment (Cohort 3 = 5 patients)
Drug: Romidepsin cycle 3 — Romidepsin administration (5mg/m²) at days 73, 80, 87
  Arms: 4 cycles of treatment (Cohort 3 = 5 patients)
Drug: Decitabine cycle 4 — Decitabine administration (5mg/m²) at days 105, 106, 107
  Arms: 4 cycles of treatment (Cohort 3 = 5 patients)
Drug: Romidepsin cycle 4 — Romidepsin administration (5mg/m²) at days 108, 115, 122
  Arms: 4 cycles of treatment (Cohort 3 = 5 patients)

SUMMARY:
The ANRS 171 SYNACTHIV trial is a monocenter pilot open label phase I trial. This trial will evaluate new procedures in LRA administration in 3 successive cohorts. In case of grade 3 to grade 5 adverse events, the inclusions and treatments will be (but not in a definitive manner) discontinued until the DSMB will conclude that the event was unrelated. Enrolment in cohort 2 then in cohort 3 will start only if no clinical grade 3 to grade 5 adverse event related to the LRAs occurs in the previous cohort.

DETAILED DESCRIPTION:
Combination antiretroviral therapy (cART) is potent but not curative. cART requires lifelong adherence. Although multiple reservoirs may exist, the HIV-1 reservoirs containing stably-integrated, transcriptionally-silent but replication-competent proviruses, are recognized to predominate among infected CD4+ T cells. They are therefore a permanent source for virus reactivation and could be responsible for the rebound of plasma viremia observed after cART interruption. Persistence of truly latent (i.e. non-defective) HIV-1 proviruses represents a major obstacle to eradication, as suggested by the failure of cART intensification strategies at clearing the viral reservoirs. Indeed, the levels of HIV-1 reservoirs appear as one of the critical factors influencing the duration of a remission after cART cessation 4. Consequently, a decline of the HIV-1 latent reservoirs size to a level sufficient to permit an efficient control of the infection by the host immune system might allow interruptions in therapy ("treatment-free windows"). Reactivation of HIV gene expression in latently-infected cells together with an efficient or intensified cART could serve as an adjuvant therapy aimed at eliminating/decreasing the pool of latent viral reservoirs.

The chromatin organization and the epigenetic control of the HIV-1 promoter are key elements involved in transcriptional silencing. The repressive nucleosome nuc-1, located immediately downstream of the transcription start site, is maintained hypoacetylated by histone deacetylases (HDACs) in latent conditions. The use of HDAC inhibitors (HDACis) as latency reversing agents (LRAs) has been well characterized in several latency models and in ex vivo cART-treated HIV-1+ patient cell cultures. Several clinical studies and trials using HDACis were reported [VPA (by Margolis, Siliciano, Lambotte and Routy), SAHA (by Margolis and by Lewin), Panobinostat (by Rasmussen) and romidepsin (by Mellors (ClinicalTrials.gov NCT01933594) and Sogaard)]. The previous studies testing VPA did not show any benefit from this HDACi in reducing the number of latently-infected resting CD4+ T cells. Two clinical trials have demonstrated that administration to cART-treated patients of a single or multiple clinically tolerable dose(s) of SAHA was temporally associated with an increase expression of cell-associated unspliced (CA-US) HIV-1 RNA levels within resting CD4+ T cells in vivo. However, both trials could neither show an increase of residual viremia nor a decrease of the size of HIV-1 reservoirs. Another recent pilot clinical trial with the HDACi Panobinostat has shown a signiﬁcant increase in CA-US RNA levels but also an increase of plasma HIV genomic RNA level analyzed by a transcription-mediated amplification (TMA) assay as well as a transient decrease in total HIV DNA level. Following cART interruption, this latter trial has shown in some patients a viral load rebound which was delayed compared to the rebound observed in most patients 2-3 weeks after stopping cART. Results from another recent pilot clinical trial including intravenous romidepsin injection, administrated once weekly for 3 weeks while maintaining cART, have shown that 5 out of 6 aviremic patients tested presented viral load levels quantifiable by standard commercial assays. Altogether, these studies are encouraging but question the efficiency of HDACi used alone to reduce the size of the HIV-1 reservoirs or to observe a delay in the viral rebound. The investigators propose some hypotheses in order to explain these partial results and some optimizations to improve therapeutic reactivation strategies:

1. The level of reactivation obtained in these clinical trials was too weak. Targeting simultaneously different mechanisms of latency should be more efficient when viral eradication is the objective since the combination of different classes of compounds could synergize (i.e. result in a higher reactivation level than the sum of the reactivations produced by each compound individually) to reactivate HIV expression in latently-infected cells.
2. A precise time schedule for LRA administration may be needed, suggesting that a sequential treatment could improve the effect of administration of two LRAs targeting different latency mechanisms.
3. HIV-1 latency is a heterogeneous phenomenon. Indeed, the investigators have previously observed in our reactivation studies performed ex vivo a high diversity among the patient cell cultures in terms of pattern of responses to the different LRAs tested. These findings suggest that HIV-1 transcriptional repression results from heterogeneous combinations of molecular mechanisms which vary from one patient to the other. The heterogeneity that the investigators have observed between patients emphasizes the need to evaluate the efficacy of an LRA first ex vivo in cell cultures from a given patient before the administration of this LRA to this given patient in vivo in the context of a clinical trial. Unfortunately, in the vast majority of the previous clinical trials aimed at reactivating HIV-1 from latency, a pre-selection based on ex vivo reactivation assays has not been performed.
4. Gene expression induction of latent HIV proviruses is stochastic. Indeed, Siliciano's group has shown that after one round of in vitro maximum T-cell activation, some proviruses remain silent but are potentially inducible after additional rounds of activation. In order to maximize the activity of a given LRA, it should thus be administered repeatedly at multiple time points.

Consequently, an optimization of the "shock" part, first part of the "shock and kill" strategy, would involve an individualized and combined treatment of LRAs, administered with a precise time schedule and repeatdly at multiple time points. In order to set up such a type of clinical trial, the investigators have investigated in vitro and ex vivo several types of LRA combination. One of them presented several advantages and was approved in human therapy.

Indeed, epigenetically, it is known that DNA methylation and histone deacetylation cooperate to establish and maintain a heterochromatin environment. Indeed, MethylBinding Domain (MBD) proteins bound to methylated DNA in cis-regulators regions can serve as bridges between DNA and chromatin-modifying factors (such as HDACs). In the case of HIV, the HIV-1 promoter has been previously shown to be hypermethylated ex vivo and resistant to reactivation in the latent reservoirs from aviremic HIV-1 infected individuals, as opposed to the hypomethylated 5'LTR of integrated proviruses present in viremic patients. Interestingly, Trejbalova et al. have very recently reported that DNA methylation of the HIV-1 promoter increases progressively during cART treatment. Indeed, these authors have detected low levels of 5' LTR DNA methylation in the resting CD4+ T cells of patients who were cART-treated for up to 3 years. However, after long-term cART, they have observed an accumulation of 5' LTR DNA methylation in the latent reservoir. The DNA methylation status of the HIV-1 promoter could contribute to "lock" the silent state of the provirus in cooperation with histone repressive posttranslational modifications such as histone deacetylation, thereby making the return of the provirus to an active state more difficult. In this view, demethylating agents could represent promising candidate drugs in combination with HDACis for reducing the pool of latent HIV reservoirs of patients under cART during at least 3 years.

Moreover, it is known that the two epigenetic modifications, DNA methylation and histone deacetylation, are dynamically linked and result in the silencing of genes in cancers. Indeed, several preclinical studies support the view that pharmacologic targeting of both DNMT and HDAC may result in synergistic anticancer activity. Moreover, two clinical trials with the DNA methylation inhibitor Decitabine and the HDACi romidepsin are ongoing in cancer therapy (NCT00037817, NCT00114257). The DNA methylation inhibitor Decitabine approved in human therapy and HDACis present several advantages for HIV-1 purging strategies. Decitabine presents the advantage to cross the blood-brain barrier, to possess an excellent distribution in body fluids, to not induce global T-cell activation. HDACis do not induce global T-cell proliferation or activation, act in a broad spectrum of cell types and potently repress CXCR4 chemokine receptor expression and function. HDACis have also been identified as new P-TEFb-releasing agents. This is undoubtedly another crucial mechanism through which HDACis reactivate HIV expression. Indeed, the switch from promoter proximal pausing to productive elongation is mediated by the viral trans-activator Tat and P-TEFb, an essential cellular elongation transcription factor. In cells, P-TEFb exists in active and inactive forms. Its release from the inactive 7SK small nuclear ribonucleoprotein complex is a critical step for P-TEFb to activate transcription elongation. Thus, importantly, the use of the two drugs might impact other mechanisms (other than histone acetylation and DNA methylation) involved in HIV latency.

1.2 Research hypothesis Recently, our laboratory has evaluated the therapeutic potential of demethylating agents in combination with HDACis in reactivating HIV from latency in vitro and ex vivo. HIV-1 reactivation potential of LRAs was assessed first in vitro in two latently-infected T-cell lines (by quantification of HIV-1 transcription, expression and production) and next ex vivo in CD8+-depleted PBMCs and resting CD4+ T-cell cultures from 58 cART-treated aviremic HIV-1+ patients (by quantification of HIV-1 production). The investigators have shown that the DNA methylation inhibitor 5-aza-2'deoxycytidine (Decitabine), but not 5-azacytidine, induced HIV expression in vitro. The investigators next demonstrated in vitro that a sequential treatment of Decitabine + HDAC is used at clinically tolerable doses synergistically induced HIV expression, highlighting for the first time the importance of a treatment schedule for LRAs combined treatments. Importantly, the investigators have shown the physiological relevance of this synergy and sequential aspect ex vivo. Interestingly, the sequential decitabine + romidepsin combinatory treatment tested induced HIV-1 recovery in a higher manner than the drugs alone in CD8+-depleted PBMCs cultures. In conclusion, the investigators reported for the first time that, in addition to the combinatory aspect, the sequential aspect of LRA administration might be critical for purging strategies aimed at decreasing the reservoir size.

The investigators hypothesize that such sequential combinatory reactivation approaches could lead to a decline in HIV-1 reservoir size to a level sufficient to allow control of the HIV infection by the host immune system and hopefully therapeutic interruptions. However, the first step in order to highlight the benefit of this type of intervention is to evaluate the feasibility, the safety and the tolerability of such sequential combinatory reactivation approaches.

Consequently, based on our ex vivo results and on our proposed optimizations of the "shock" part, first part of the "shock and kill" strategy, (involving an individualized and combined treatment of LRAs, administered with a precise time schedule and repeatedly at multiple time points), the investigators propose to set up a phase I trial in HIV-1 sub-type B positive patients under cART for at least 48 months and presenting, to the best knowledge of the clinical PI, no detectable viral blip for at least 12 months in order to evaluate the feasibility, safety and tolerability of a sequential treatment of Decitabine in combination with romidepsin delivered at multiple time points [one time (cohort 1), two times (cohort 2) or four times (cohort 3)]. As a secondary objective, the investigators will also evaluate the impact on viral reservoirs and HIV gene expression of the combinatory treatment (decitabine + romidepsin).

ELIGIBILITY:
Inclusion Criteria:

* Man aged 18-69 years;
* Man with documented infection with sub-type B HIV-1;
* On cART since more than 36 months before pre- screening and at a stable regimen for at least 2 months before pre-screening and until inclusion;
* HIV plasma viral load persistently < the threshold (of the local test used) and undetectable during the 12 months prior to pre-screening and until inclusion;
* CD4+ T-cells count nadir ≥ 200 cells per mm3 documented in the medical file; Transient CD4+ T-cells count < 200 cells per mm3 is allowed for a short period if the value is associated with a single isolated acute infection
* CD4+ T-cells count ≥ 500 cells per mm3 for at least 12 months before pre-screening and until inclusion;
* EBV viral load < 1000 cp.mL-1, CMV viral load < 10000 cp mL-1;
* Able and willing to comply with study visits and procedures as per protocol;
* Able to understand, sign and date the written voluntary informed consent form at the pre screening visit prior to any protocol-specific procedures.
* Free, informed and written consent signed by the person and the investigator (at the latest on the day of pre-screening and before any investigation carried out as part of the trial) (law of 7 May 2004. article 6)

Exclusion Criteria:

* Man who want to father a child or refuse contraception (condoms) while receiving treatment and for 3 months following completion of treatment; Man with a female partner of childbearing potential who refuses to use a highly effective contraceptive method during the same period (Experimental treatment period and for 3 months following completion of experimental treatment).
* Clinically significant cardiac disease including QTc-prolongation (QTc value > 450msec);
* On PI based regimen or regimen containing NNRTI (except Doravirine which is allowed), Ritonavir or Cobicistat;
* Treated with CYP 450 inducer or inhibitor, in particular dexamethasone, carbamazepine, phenytoin, rifabutin, rifapentine and phenobarbital;
* Treated with anti-arrhythmic medicines or medicinal products that lead to significant QT prolongation;
* Treated with warfarin or coumarin derivative;
* History of an AIDS-defining clinical illness (based on CDC classification);
* Active coinfection with viral hepatitis B;
* Active coinfection with viral hepatitis C;
* Received any vaccination within 4 weeks prior to the first administration of the study products and plan to receive throughout the study (with the exception of influenza and COVID-19 vaccines which can be injected 4 weeks after the last administration of the study products as well as the Monkeypox vaccination that will be allowed during trial if participant becomes a contact at risk for monkeypox infection (according to national recommendations));
* Treated with sexual hormone during the administration period of the study treatments (until CXD32);
* Active malignancy that may require chemotherapy or radiation therapy;
* Any significant acute medical illness in the 8 weeks prior to pre-screening and until inclusion;
* Haematological or biochemical laboratory parameters at pre-screening and screening : Hemoglobin (<LLN), absolute neutrophil count (<LLN), platelets (<LLN), INR (>1.2), Partial Thromboplastin Time (>ULN); grade ≥ 2 for the following parameters: Total serum Creatinine, urea, uric acid, glycemia, total serum bilirubin, Alkaline Phosphatase (ALP) AST-ALT, gammaglutamyl transferase (GGT), lipasemia, LDH, Ionogram: Na, K, Ca, Mg, CRP, albumin, proteins, CPK;
* Liver insufficiency (Child Pugh score >5);
* Kidney insufficiency (Estimation of glomerular filtration<60mL/mn/1,73m2 ; evaluation with CKDepi formula, according to the 2012 French Haute autorité de santé recommandations);
* Participant under guardianship or curatorship or deprived of their liberty by a judicial or administrative decision
* Participant potentially inable to follow the protocol requirements (e.g. comprehension of the study requirements, ability to understand and comply with procedures for collection of safety data, expressed availability for the required study period, and ability and willingness to attend scheduled visits).
* Participating to another interventional study or still in an exclusion period from another clinical trial ;
* Planning to participate in a study within 3 months after the end of the present trial.

Ages: 18 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events (SAE) and severe clinical or biological adverse events (AE) related to the study drugs | within 2 weeks after the last injection for each patient
  Incidence of Serious Adverse Events (SAE) and severe clinical or biological adverse events (AE) related to the study drugs, , according to CTCAE scale, per patient

SECONDARY OUTCOMES:
Incidence of clinical and biological adverse events (AE) of all grades | through study completion, an average of 4 years
  Incidence, severity and relation to study products of clinical and biological adverse events (AE) of all grades according to CTCAE scale, per cohort
Efficacy of the treatment on the HIV reservoir | At pre-screening, before the first dose of each cycle (day 1), 1 hour following each romidepsine administration (day 4, day 11, day 18), at the end of each cycle (day 32), at each follow-up visit (Follow-up days 28, 84, 140, 364) of each cohort.
  Number of total HIV-1 DNA log copies /10e6 cells by an ultrasensitive assay
Blood concentration of decitabine and romidepsin after injection | day 1, day 4, day 11; day 18 of cycle 1
  The blood concentration of decitabine and romidepsin after injection. HPLC will be performed on plasma samples collected 5 minutes before the end of drug's administration
Capacity of latently-infected cells to be reactivated | at pre-screening, at day 32 of each cycle of treatment, at follow-up visit day 140 of each cohort
  capacity of latently-infected cells to be reactivated, by the decitabine+romidepsin combination assessed by ex vivo reactivation assay
Increase in viral load | at pre-screening and at day 1 of each cycle (prior decitabin treatment), day 25 and day 32, and at each follow-up visit ((day 28, day 84, day 140, day 364)
  Increase in viral load assessed by the classical method performed by the patient's hospital with a threshold at 20 copies/mL or 40 copies/mL
Increase in viral load | at pre-screening, day 1 on each cycle (prior decitabin treatment), 1 hour following each romidepsine administration (day 4, day 11, day 18), at the end of each cycle (day 32), and at each follow up visits (day 28, day 84, day 140, day 364)
  Increase in viral load assessed by an ultrasensitive method with a threshold at 5-10 copies/ml or <2 copies/ml
HIV-1 transcripts measure | at pre-screening, day 1, day 4, day 11, day 18, day 32.
  The HIV-1 transcripts by an ultrasensitive assay

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Saint-Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Research projects may be submitted and evaluated by the Trial Scientific committee for scientific relevance. If the projects receives a favorable opinion, a data sharing agreement shall be signed.
  Participants will be informed of any further research project and will have the opportunity to refuse the use of their data